CLINICAL TRIAL: NCT00001500
Title: Genetic Factors and Interrelationships for Cancer Risk-Related Behaviors and Complex Traits
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960061; 96-C-0061
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-07

CONDITIONS: Acquired Immunodeficiency Syndrome; Alcoholism; HIV Infection; Neoplasm; Smoking
Keywords: Smoking; Alcohol; HIV; AIDS; DNA Markers; Personality; Healthy Volunteers; Normal Volunteer
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Alcoholism; HIV Infections; Neoplasms; Smoking

SUMMARY:
We propose to conduct a multifactorial genetic study of cancer risk-related behaviors and other complex human characteristics. The main areas of interest are tobacco smoking, excess alcohol consumption, psychological traits, and HIV/AIDS susceptibility and progression. The subjects will be adult male and female probands who display one or more of the phenotypes of interest together with their brothers, sisters and parents. Information on tobacco and alcohol use, psychological and personality traits, sexual behavior, HIV status and progression, and other characteristics with possible genetic components will be obtained through structured interviews and questionnaires. DNA will be prepared from blood samples and typed for a series of candidate genes chosen for function and for random polymorphic markers. By correlating the genotypic and phenotypic information, we hope to identify individual loci that interactively contribute to many different aspects of human health and disease.

DETAILED DESCRIPTION:
We propose to conduct a multifactorial genetic study of cancer risk-related behaviors and other complex human characteristics. The main areas of interest are tobacco smoking, excess alcohol consumption, psychological traits, and HIV/AIDS susceptibility and progression. The subjects will be adult male and female probands who display one or more of the phenotypes of interest together with their brothers, sisters and parents. Information on tobacco and alcohol use, psychological and personality traits, sexual behavior, HIV status and progression, and other characteristics with possible genetic components will be obtained through structured interviews and questionnaires. DNA will be prepared from blood samples and typed for a series of candidate genes chosen for function and for random polymorphic markers. By correlating the genotypic and phenotypic information, we hope to identify individual loci that interactively contribute to many different aspects of human health and disease.

ELIGIBILITY:
INCLUSION CRITERIA:

The basic requirement for entry in the study will be the presence of any individual smoker who is willing to complete the evaluation process and donate a blood sample.

Additional siblings will be encouraged but not required to participate.

Probands will be recruited through smoking cessation programs at the National Naval Medical Center.

Attendees at programs offered by the Health Promotions Department and the Military Family Health Center will be invited to participate in this study.

EXCLUSION CRITERIA:

All subjects will be adults (greater than 18 years).

There will be no exclusions based on sex, ethnic group, or race.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4500
Dates: Start 1996-04; Study Completion 2004-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Carmelli D, Swan GE, Robinette D, Fabsitz RR. Heritability of substance use in the NAS-NRC Twin Registry. Acta Genet Med Gemellol (Roma). 1990;39(1):91-8. doi: 10.1017/s0001566000005602. PMID 2392895
- [Background] Carmelli D, Swan GE, Robinette D, Fabsitz R. Genetic influence on smoking--a study of male twins. N Engl J Med. 1992 Sep 17;327(12):829-33. doi: 10.1056/NEJM199209173271201. PMID 1508241
- [Background] Swan GE, Carmelli D, Rosenman RH, Fabsitz RR, Christian JC. Smoking and alcohol consumption in adult male twins: genetic heritability and shared environmental influences. J Subst Abuse. 1990;2(1):39-50. doi: 10.1016/s0899-3289(05)80044-6. PMID 2136102